CLINICAL TRIAL: NCT00726869
Title: A Phase 1/2, Multi-center, Open-label, Dose-escalation Study of Elotuzumab(Humanized Anti-CS1 Monoclonal IgG1 Antibody) and Bortezomib in Subjects With Multiple Myeloma Following One to Three Prior Therapies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment has been halted
Sponsor: Abbott (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HuLuc63-1702
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Myeloma
Keywords: Patients After One to three Prior Therapies
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 2.5 mg/kg
  Interventions: Drug: Elotuzumab (HuLuc63)
- Cohort 2 (Experimental): 5.0 mg/kg
  Interventions: Drug: Elotuzumab (HuLuc63)
- Cohort 3 (Experimental): 10.0 mg/kg
  Interventions: Drug: Elotuzumab (HuLuc63)
- Cohort 4 (Experimental): 20.0 mg/kg
  Interventions: Drug: Elotuzumab (HuLuc63)

INTERVENTIONS:
Drug: Elotuzumab (HuLuc63) — Cohort 1 - 2.5 mg/kg elotuzumab IV with bortezomib on Days 1 & 11, with only Bortezomib IV on Days 4 & 8; Cohort 2 - 5.0 mg/kg elotuzumab IV with bortezomib on Days 1 & 11, with only Bortezomib IV on Days 4 & 8; Cohort 3 - 10.0 mg/kg elotuzumab IV withbortezomib on Days 1 & 11, with only Bortezomib IV on Days 4 & 8; and Cohort 4 - 20.0 mg/kg elotuzumab IV with bortezomib on Days 1 & 11, with only Bortezomib IV on Days 4 & 8.
  Other Names: Elotuzumab

SUMMARY:
This Phase 1/2, multi-center, open-label, multiple-dose, dose escalation study will evaluate the combination of elotuzumab and bortezomib in subjects with MM following 1 to 3 prior therapies. For the Phase 1 portion, elotuzumab will be administered by intravenous (IV) infusion at up to 4 dose levels ranging from 2.5 mg/kg to 20.0 mg/kg within 30 minutes following the administration of bortezomib at 1.3 mg/m^2 IV bolus. Bortezomib will be given in 21 day cycles (twice weekly for 2 weeks on Days 1, 4, 8, and 11 followed by a 10-day rest period). Elotuzumab will be administered as a separate infusion within 30 minutes following bortezomib administration on the same days as the first and last dose of each bortezomib cycle (i.e., Days 1 and 11).

DETAILED DESCRIPTION:
The phase 2 portion of this study was not initiated because a decision was made to conduct a phase 2 randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria

1. Males or females, age 18 years or older.
2. Diagnosis of MM and documentation of 1 to 3 prior therapies.
3. M-protein spike (complete immunoglobulin molecule) of >= 1g/dL in serum and/or >= 0.5 g excreted in a 24-hour urine collection sample. Light chain only disease is not an inclusion criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. No prior bortezomib treatment OR responsive (PR or better) to prior bortezomib treatment for a minimum of 3 months OR responsive to prior bortezomib treatment at the time of going to another treatment or ceasing treatment.
6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <=3 x upper limit of normal (ULN).
7. Total bilirubin <=2 x ULN.
8. Serum creatinine <=2.0 mg/dL (unless related to MM, then <=3.0 mg/dL).
9. Must have adequate bone marrow function defined as:

   * Absolute neutrophil count >1,000 cells/mm3 (1.0 x 10^9 cells/L) without growth factor support for 7 days;
   * Platelets >=75,000 cells/mm3 (75 x 10^9 cells/L) without transfusion within 72 hours of screening;
   * Hemoglobin >=8 g/dL without red blood cell transfusion within 2 weeks of screening;
10. Serum calcium (corrected for albumin) level at or below ULN range (treatment of hypercalcemia is allowed and subject may enroll if hypercalcemia returns to normal with standard treatment); additional screening time may be allowed for confirmation - consult with sponsor's medical monitor.
11. Use of appropriate contraception where applicable.
12. Negative urine pregnancy test where applicable.
13. Must have 2-dimensional echocardiogram indicating left ventricular ejection fraction (LVEF) >=45% within 30 days prior to the first dose of elotuzumab.
14. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Exclusion Criteria

1. Life expectancy of less than 3 months.
2. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years.
3. Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary,(including acute diffuse infiltrative pulmonary and pericardial disease), hepatic, and renal diseases unless renal insufficiency is felt to be secondary to MM.
4. Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
5. Prior treatment with bortezomib in 3 months prior to the first dose.
6. Thalidomide, lenalidomide cytotoxic chemotherapy, or corticosteroids (except prior to infusion of first dose of study drug as prophylaxis for infusion reactions) within 2 weeks of the first dose of elotuzumab.
7. Prior therapy with anti-CD56+ therapeutics.
8. Radiotherapy within 2 weeks prior to the first dose of elotuzumab.
9. Investigational drug within 3 weeks or 3x the half-life of the investigational drug (whichever is longer ) of the first dose of elotuzumab.
10. Prior peripheral stem cell transplant within 12 weeks of the first dose of elotuzumab.
11. Nitrogen mustard agents, melphalan, or monoclonal antibodies within 6 weeks of the first dose of elotuzumab.
12. Neuropathy >=Grade 2 (NCI CTCAE v3.0).
13. Current orthostatic hypotension.
14. Known active infections requiring antibiotic, antiviral, or antifungal therapy.
15. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation.
16. Any condition that in the investigator's opinion makes the subject unsuitable for study participation.
17. Hypersensitivity to recombinant proteins or excipients in elotuzumab or bortezomib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Identify the maximum tolerated dose of elotuzumab in combination with bortezomib (phase 1). | First cycle of treatment.
  The highest dose level of elotuzumab at which <= 1 dose-limiting toxicity occurs in 6 subjects
Evaluate the efficacy of elotuzumab in combination with bortezomib (phase 2). | Screening to the 30 day follow up visit.
  Objective response rate (complete and partial response) according to European Group for Blood and Marrow Transplantation (EBMT) criteria

SECONDARY OUTCOMES:
Evaluate the efficacy of elotuzumab in combination with bortezomib (phase 1). | Screening to the 30 day follow up visit.
  Objective response rate according to EBMT criteria, duration of response, time to progression, and progression-free survival
Evaluate the safety of elotuzumab in combination with bortezomib (phase 1 and 2). | Screening to the 30 day follow up visit.
  Frequency, severity, and relationship of adverse events and serious adverse events with the combination of elotuzumab and bortezomib
Evaluate the pharmacokinetic parameters of elotuzumab in combination with bortezomib (phase 1 and 2) | Screening to the 30 day follow up visit.
  Pharmacokinetic profile
Evaluate the immunogenicity of elotuzumab in combination with bortezomib (phase 1 and 2). | Screening to the 30 day follow up visit.
  Incidence of elotuzumab-specific antidrug antibodies
Evaluate the pharmacodynamics of elotuzumab in combination with bortezomib (phase 1 and 2). | Screening to the 30 day follow up visit.
  Changes in pharmacodynamic endpoints as they relate to dose, response, and toxicity of elotuzumab in combination with bortezomib

CONTACTS AND LOCATIONS:
Overall Officials: Anil Singhal, PhD, Study Director — Abbott
Locations (8):
- United States (8):
  - Site Reference ID/Investigator# 63853, Los Angeles, California
  - Site Reference ID/Investigator# 63855, Chicago, Illinois
  - Site Reference ID/Investigator# 63847, Boston, Massachusetts
  - Site Reference ID/Investigator# 63852, Ann Arbor, Michigan
  - Site Reference ID/Investigator# 63854, Hackensack, New Jersey
  - Site Reference ID/Investigator# 63850, Buffalo, New York
  - Site Reference ID/Investigator# 63849, Columbus, Ohio
  - Site Reference ID/Investigator# 63848, Seattle, Washington